CLINICAL TRIAL: NCT07303530
Title: Effect of Printing Layer Thickness on Growth of Candida Albicans in Completely Edentulous Patients Rehabilitated With 3D-Printed Maxillary Complete Denture Bases: A Randomized Cross-over Study
Brief Title: Effect of Printing Layer Thickness on Growth of Candida Albicans in Completely Edentulous Patients Rehabilitated With 3D-Printed Maxillary Complete Denture Bases.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed abdelgawad mousa, assistant lecturer "principal investigator", Cairo University
Allocation: Not Applicable | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 3354445
Record Dates: First submitted 2025-11-25; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Printed Dentures
Keywords: Candida
MeSH Terms: conditions — Torulopsis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: printing layer thickness of denture — denture printed by multiple printing layer thicknesses to assess effect of layer thickness on fungal growth
  Other Names: other printing layer thickness

SUMMARY:
In completely edentulous patients rehabilitated with 3D-printed maxillary dentures bases, does the printing layer thickness affect candidal adherence and growth on the fitting surface of dentures.

DETAILED DESCRIPTION:
The trial will follow a cross-over design, where each participant will wear denture bases printed with three different layer thicknesses (25 µm, 50 µm, and 100 µm) at a random order. Each participant will wear each of the three dentures for an 8-week period, with a washout period of two weeks between each thickness.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients aged 30-80 years
* Oral cavity is free from any mucosal lesions.
* No systemic conditions that would contraindicate participation in the study.

Exclusion Criteria:

* History of allergic reactions to denture materials.
* Active mucosal lesions related to denture use.
* Pregnancy or lactation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-12-05 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Candidal growth | 8-10 weeks
  candidal growth over denture surface measured by colony-forming units (CFU)

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - cairo University hospital, Cairo, Cairo Governorate
  - faculty of dentistry Cairo hospital, Cairo, Cairo Governorate